CLINICAL TRIAL: NCT01982955
Title: A Phase Ib/II Multicenter, Randomized, Open Label Trial to Compare Tepotinib (MSC2156119J) Combined With Gefitinib Versus Chemotherapy as Second-Line Treatment in Subjects With MET Positive, Locally Advanced or Metastatic NSCLC Harboring EGFR Mutation and Having Acquired Resistance to Prior EGFR-TKI Therapy (INSIGHT)
Brief Title: Tepotinib With Gefitinib in Participants With Locally Advanced or Metastatic NSCLC (INSIGHT)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200095-006; 2016-001604-28 (EudraCT Number)
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: MSC2156119J; Gefitinib; Pemetrexed; Cisplatin; MET positive; Tepotinib; Carboplatin; INSIGHT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tepotinib; Gefitinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg (Experimental): Participants received Tepotinib 300 milligram (mg) along with 250 mg Gefitinib tablets orally once daily over a 21-day treatment cycle until progressive disease, intolerable toxicity or withdrawal from treatment.
  Interventions: Drug: Tepotinib; Drug: Gefitinib
- Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg (Experimental): Participants received Tepotinib 500 milligram (mg) along with 250 mg Gefitinib tablets orally once daily over a 21-day treatment cycle until progressive disease, intolerable toxicity or withdrawal from treatment.
  Interventions: Drug: Tepotinib; Drug: Gefitinib
- Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 negative) (Experimental): Participants randomized to receive Tepotinib recommended Phase 2 dose 500 mg once daily along with 250 mg Gefitinib tablets orally once daily over a 21-day cycle until progressive disease, intolerable toxicity or withdrawal from treatment.
  Interventions: Drug: Tepotinib; Drug: Gefitinib
- Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 negative) (Experimental): Participants randomized to receive 500 milligram per square meter (mg/m^2) of Pemetrexed as intravenous infusion over 10 minutes in combination with Cisplatin (75 mg/m2 as an intravenous infusion over 2 hours) or Carboplatin (intravenously at a dose of area under curve (AUC) 5 or AUC6 at the discretion of the Investigator) on Day 1 of each 21-day cycle until progressive disease, intolerable toxicity or withdrawal from treatment or up to 6 cycles if or 4 cycles followed by Pemetrexed maintenance monotherapy.
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Phase 2: Single-arm Cohort (MET+ T790M positive) (Experimental): Participants with MET+ T790M positive Non-small Cell Lung Cancer (NSCLC) received a Tepotinib recommended Phase 2 dose 500 mg once daily along with 250 mg Gefitinib tablets orally once daily over a 21-day treatment cycle until progressive disease, intolerable toxicity or withdrawal from treatment.
  Interventions: Drug: Tepotinib; Drug: Gefitinib

INTERVENTIONS:
Drug: Tepotinib — Tepotinib was administered at a dose range of 300 or 500 milligram (mg) (Phase 1b) and the recommended phase II dose (RP2D) determined in the Phase 1b in Phase II orally once daily over a 21-day cycle until progressive disease, intolerable toxicity, participants withdrawal from treatment. RP2D was determined as per safety monitoring committee (SMC) discretion.
  Arms: Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg; Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg; Phase 2: Single-arm Cohort (MET+ T790M positive); Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 negative)
Drug: Gefitinib — Gefitinib was administered at a dose of 250 mg orally as once daily over a 21-day cycle until progressive disease, intolerable toxicity, participants withdrawal from treatment.
  Arms: Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg; Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg; Phase 2: Single-arm Cohort (MET+ T790M positive); Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 negative)
Drug: Pemetrexed — Pemetrexed was administered at a dose of 500 milligram per square meter (mg/m^2) as intravenous infusion over 10 minutes on Day 1 of each 21-day cycle until progressive disease, intolerable toxicity, participants withdrawal from treatment or up to 6 cycles if pemetrexed maintenance is not considered.
  Arms: Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 negative)
Drug: Cisplatin — Cisplatin was administered at a dose of 75 mg/m^2 as intravenous infusion over 2 hours on Day 1 of each 21-day cycle until progressive disease, intolerable toxicity, participants withdrawal from treatment or up to 6 cycles if pemetrexed maintenance is not considered.
  Arms: Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 negative)
Drug: Carboplatin — Carboplatin was administered intravenously on Day 1 of each 21-day cycle at a dose of area under curve (AUC) 5 or AUC6 at the discretion of the Investigator until progressive disease, intolerable toxicity, participants withdrawal from treatment or up to 6 cycles if pemetrexed maintenance is not considered.
  Arms: Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 negative)

SUMMARY:
This is a multi-center, open-label, randomized, Phase 1b/2 study to determine the recommended phase 2 dose (RP2D) and to evaluate the efficacy in terms of progression free survival (PFS) of Tepotinib when used in combination with gefitinib in partcipants with T790M negative, MET positive locally advanced or metastatic non-small cell lung cancer (NSCLC) harboring epidermal growth factor receptor (EGFR) mutation and having acquired resistance to Prior EGFR-Tyrosine Kinase Inhibitor (EGFR-TKI) Therapy. This study has 2:1 randomization (Tepotinib/Gefitinib arm versus Chemotherapy arm).

ELIGIBILITY:
Phase Ib

Inclusion Criteria:

* Histologically or cytologically confirmed advanced non-small cell lung cancer (NSCLC), regardless of histology subtype, which failed on gefitinib for reasons other than toxicity or compliance;
* Availability of a fresh or archived pre treatment tumor biopsy (excluding fine needle aspiration and cytology samples). For participants who have had at least 1 prior anticancer treatment, a biopsy obtained between failure of the most recent anticancer treatment and enrolment is mandatory;
* Mesenchymal-epithelial transition diagnostic-positive (status) (MET+ status), as determined by the central laboratory
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Other protocol defined inclusion criteria could apply.

Phase II

Inclusion criteria:

* Locally advanced or metastatic NSCLC other than predominantly squamous histology (confirmed by either histology or cytology);
* Activating mutation of the epidermal growth factor (EGFR) receptor (documented, or as determined by the central laboratory)
* Acquired resistance on first-line EGFR-Tyrosine Kinase Inhibitors (EGFR-TKI) therapy including gefitinib, erlotinib, icotinib, or afatinib
* EGFR T790M status after acquired resistance to first line EGFR-TKI therapy including gefitinib, erlotinib, icotinib, or afatinib treatment (as determined by the central laboratory, using a validated PCR test);
* T790M negative status for the randomized part
* T790M positive status for the single-arm cohort (mainland China sites only)
* Availability of a fresh or archived tumor tissue (excluding fine needle aspiration and cytology samples) obtained between documentation of acquired resistance to gefitinib, erlotinib, icotinib, or afatinib and enrollment is mandatory
* MET+ status, as determined by the central laboratory i.e. c-Met overexpression as determined by IHC (i.e., IHC 2+ or IHC 3+) and/or c-Met amplification and/or increased c-Met gene copy number (GCN), both determined by ISH;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria (Phase I and II):

* Estimated life expectancy less than (<) 3 months
* Inadequate bone marrow, liver or renal functions
* Prior chemotherapy, biological therapy, radiation therapy, or other investigational anticancer therapy (not including palliative radiotherapy at focal sites) within 21 days prior to the first dose of study treatment (Phase 1b only)
* Prior systemic anticancer treatment with chemotherapy or other agents targeting the EGFR pathway excluding gefitinib, erlotinib, icotinib, and afatinib for advanced NSCLC (one course of chemotherapy regimen for [neo] adjuvant purpose, or one course of chemoradiation for Stage IIIa disease is allowed) (Phase 2 only)
* Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-12-23 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2021-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (44):
- China (13):
  - Beijing Cancer Hospital, Beijing
  - Beijing Chest Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Jilin University, Changchun
  - Fuzhou General Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sir Run Run Shaw Hospital Cardiology, Hangzhou
  - The First Affiliated Hospital of College of Medicine, Hangzhou
  - Shanghai Chest Hospital, Shanghai
  - Tongji Hospital, Wuhan
  - Fourth Military Medical University, Xi'an
  - Zhejiang Cancer Hospital, Zhejiang
- Italy (2):
  - Azienda Ospedaliero Universitaria Mater Domini-Campus Universitario, Catanzaro
  - IEO Istituto Europeo di Oncologia, Milan
- Malaysia (2):
  - University Malaya Medical Centre, Kuala Lumpur
  - Beacon International Specialist Centre Sdn Bhd, Petaling Jaya
- Singapore (3):
  - National Cancer Center, Singapore
  - National University Hospital, Singapore
  - Raffles Hospital, Singapore
- South Korea (13):
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Hospital, Daegu
  - Chonnam National University Hwasun Hospital, Hwasun
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Severance Hospital Yonsei University Health System, Seongnam-si
  - Asan medical Centre, Seoul
  - Gangnam Severance Hospital Yonsei University, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National Universtiy Hospital, Seoul
  - The Catholic University of Korea St Mary s Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico Universitario, Valencia
  - Hospital Alvaro Cunqueiro, Vigo
- Taiwan (7):
  - Chang Gung Memorial Hospital-Kaohsiung, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou, Taoyuan District

REFERENCES:
- [Result] Wu YL, Cheng Y, Zhou J, Lu S, Zhang Y, Zhao J, Kim DW, Soo RA, Kim SW, Pan H, Chen YM, Chian CF, Liu X, Tan DSW, Bruns R, Straub J, Johne A, Scheele J, Park K, Yang JC; INSIGHT Investigators. Tepotinib plus gefitinib in patients with EGFR-mutant non-small-cell lung cancer with MET overexpression or MET amplification and acquired resistance to previous EGFR inhibitor (INSIGHT study): an open-label, phase 1b/2, multicentre, randomised trial. Lancet Respir Med. 2020 Nov;8(11):1132-1143. doi: 10.1016/S2213-2600(20)30154-5. Epub 2020 May 29. PMID 32479794
- See also: Trial Awareness and Transparency website — https://clinicaltrials.merckgroup.com/en/trial-details/?id=EMR%20200095-006
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18 participants were enrolled in Phase 1b part of the study and a total of 70 participants were enrolled in phase 2 part of the study. Participants enrolled in phase 1b were not eligible for randomization in phase 2.
Groups:
- Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative): Participants randomized to receive 500 milligram per square meter (mg/m^2) of Pemetrexed as intravenous infusion over 10 minutes in combination with Cisplatin (75 mg/m^2 as an intravenous infusion over 2 hours) or Carboplatin (intravenously at a dose of area under curve (AUC) 5 or AUC6 at the discretion of the Investigator) on Day 1 of each 21-day cycle until progressive disease, intolerable toxicity or withdrawal from treatment or up to 6 cycles if or 4 cycles followed by Pemetrexed maintenance monotherapy.
Period: Overall Study
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Started | 6 | 12 | 31 | 24 | 15
Treated | 6 | 12 | 31 | 23 | 15
Completed | 6 | 12 | 31 | 23 | 15
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Randomized but not treated | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive) | Total
Number analyzed (Participants) | 6 | 12 | 31 | 24 | 15 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 21 | 17 | 9 | 56
  >=65 years | 3 | 6 | 10 | 7 | 6 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 20 | 12 | 10 | 52
  Male | 3 | 5 | 11 | 12 | 5 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 12 | 31 | 24 | 15 | 88
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants Experiencing at Least One Dose Limiting Toxicity (DLT)
Description: Dose limiting toxicity (DLT) using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.0 was defined as toxicities at any dose level and judged to be related to the study treatment by investigator and/or the sponsor. DLTs included Grade 4 neutropenia for more than 7 days; Grade greater than or equal to (>=) 3 febrile neutropenia for more than 1 day; Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with non-traumatic bleeding; Grade >= 3 uncontrolled nausea/vomiting and/or diarrhea despite adequate and optimal treatment and Grade >= 3 any non-hematological adverse event (AE), except the aforementioned gastrointestinal events and alopecia. Number of participants who experienced DLT during Phase 1b were reported.
Time Frame: Day 1 to Day 21 of Cycle 1 (each cycle is 21 days)
Population: Dose Limiting Toxicity (DLT) set included all participants who experienced a DLT during Cycle 1, or received at least 80 percent of all planned doses of treatment during Cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 3 | 12
Participants | 0 | 0

2. Primary Outcome: Phase 1b: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs include both Serious TEAEs and non-serious TEAEs. Number of Participants with TEAEs and serious TEAEs were reported.
Time Frame: Up to 175 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Participants
  Any TEAEs | 6 | 12
  Any Serious TEAEs | 4 | 7

3. Primary Outcome: Phase 2 (Randomized Part Only): Progression-free Survival (PFS) Based on Tumor Assessment by the Investigator
Description: Progression-free survival (assessed by the Investigator) time was defined as the time in months from randomization to either first observation of radiologically confirmed progression disease (PD) by the investigator or occurrence of death due to any cause within 84 days of either randomization or the last tumor assessment. PD is defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 millimeter (mm). PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Up to 328 weeks
Population: The Intent-to-treat analysis set in the Phase 2 part of the study included all participants with treatment group who were randomized to study treatment.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative)
Number analyzed (Participants) | 31 | 24
Months | 4.86 [3.88 to 6.87] | 4.37 [4.17 to 6.80]

4. Secondary Outcome: Phase 1b: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Sampling Time AUC (0-t) of Tepotinib, Its Metabolites and Gefitinib
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration is at or above the lower limit of quantification (LLLQ). AUC(0-t) was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 1 and 15 of Cycle 1 (each Cycle is 21 days)
Population: The Pharmacokinetic (PK) set included all participants who had received at least 1 dose of the tepotinib or gefitinib and who had provided at least 1 plasma concentration measurement of tepotinib or gefitinib after the first dose. Here "Number Analyzed" signifies those participants who were evaluable for specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
nanogram*hour per milliliter (ng*h/mL)
  Tepotinib: Day 1 of Cycle 1: number analyzed (Participants) | 5 | 12
  Tepotinib: Day 1 of Cycle 1 | 6280 (25.4) | 9210 (48.4)
  Tepotinib: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 9
  Tepotinib: Day 15 of Cycle 1 | 15600 (19.6) | 22200 (43.3)
  MSC2571109A: Day 1 of Cycle 1: number analyzed (Participants) | 5 | 11
  MSC2571109A: Day 1 of Cycle 1 | 1680 (11.8) | 1770 (56.7)
  MSC2571109A Day15 of Cycle 1: number analyzed (Participants) | 6 | 8
  MSC2571109A Day15 of Cycle 1 | 4420 (25.7) | 7530 (52.6)
  MSC2571107A Day 1 of Cycle 1: number analyzed (Participants) | 5 | 11
  MSC2571107A Day 1 of Cycle 1 | 248 (49.3) | 324 (57.3)
  MSC2571107A Day 15 of Cycle 1: number analyzed (Participants) | 6 | 8
  MSC2571107A Day 15 of Cycle 1 | 872 (38.5) | 1880 (76.0)
  Gefitinib: Day 1 of Cycle 1: number analyzed (Participants) | 2 | 11
  Gefitinib: Day 1 of Cycle 1 | NA (NA) — Only 2 participants had evaluable AUC(0-t) at time point. For statistical reasons, calculation of summary statistics does not make sense for this low sample size. Individual values were 3830 and 3980 ng*h/mL. | 2930 (45.8)
  Gefitinib: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 9
  Gefitinib: Day 15 of Cycle 1 | 7690 (44.1) | 7080 (29.0)

5. Secondary Outcome: Phase 1b: Area Under the Plasma Concentration-Time Curve Within 1 Dosing Interval (AUC 0-tau) of Tepotinib, Its Metabolites and Gefitinib
Description: AUC (0-tau) is the area under the plasma concentration time curve within 1 dosing interval.
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 1 and 15 of Cycle 1 (each Cycle is 21 days)
Population: The PK set included all participants who had received at least 1 dose of the tepotinib or gefitinib and who had provided at least 1 plasma concentration measurement of tepotinib or gefitinib after the first dose. Here "Number Analyzed" signifies those participants who were evaluable for specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
ng*h/mL
  Tepotinib: Day 1 of Cycle 1: number analyzed (Participants) | 5 | 12
  Tepotinib: Day 1 of Cycle 1 | 6280 (25.4) | 9210 (48.4)
  Tepotinib: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 9
  Tepotinib: Day 15 of Cycle 1 | 15600 (19.6) | 22200 (43.3)
  MSC2571109A: Day 1 of Cycle 1: number analyzed (Participants) | 5 | 11
  MSC2571109A: Day 1 of Cycle 1 | 1680 (11.8) | 1770 (56.7)
  MSC2571109A: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 8
  MSC2571109A: Day 15 of Cycle 1 | 4420 (25.7) | 7530 (52.6)
  MSC2571107A: Day 1 of Cycle 1: number analyzed (Participants) | 5 | 11
  MSC2571107A: Day 1 of Cycle 1 | 248 (49.3) | 324 (57.3)
  MSC2571107A: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 8
  MSC2571107A: Day 15 of Cycle 1 | 872 (38.5) | 1880 (76.0)
  Gefitinib: Day 1 of Cycle 1: number analyzed (Participants) | 2 | 11
  Gefitinib: Day 1 of Cycle 1 | NA (NA) — Only 2 participants had evaluable AUC(0-tau) at time point. For statistical reasons, calculation of summary statistics does not make sense for this low sample size. Individual values were 3830 and 3980 ng*h/mL. | 2930 (45.8)
  Gefitinib: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 9
  Gefitinib: Day 15 of Cycle 1 | 7690 (44.1) | 7080 (29.0)

6. Secondary Outcome: Phase 1b: Maximum Observed Plasma Concentration (Cmax) of Tepotinib, Its Metabolites and Gefitinib
Description: Cmax is the maximum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 1 and 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per Milliliter (ng/mL)
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Nanogram per Milliliter (ng/mL)
  Tepotinib: Day 1 of Cycle 1: number analyzed (Participants) | 5 | 12
  Tepotinib: Day 1 of Cycle 1 | 375 (30.4) | 575 (62.6)
  Tepotinib: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 10
  Tepotinib: Day 15 of Cycle 1 | 763 (22.0) | 1050 (44.1)
  MSC2571109A: Day 1 of Cycle 1: number analyzed (Participants) | 5 | 11
  MSC2571109A: Day 1 of Cycle 1 | 132 (14.7) | 149 (56.5)
  MSC2571109A: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 9
  MSC2571109A: Day 15 of Cycle 1 | 280 (32.0) | 444 (45.8)
  MSC2571107A: Day 1 of Cycle 1: number analyzed (Participants) | 5 | 11
  MSC2571107A: Day 1 of Cycle 1 | 16.8 (56.5) | 24.3 (62.5)
  MSC2571107A: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 9
  MSC2571107A: Day 15 of Cycle 1 | 44.9 (40.5) | 94.9 (70.8)
  Gefitinib: Day 1 of Cycle 1: number analyzed (Participants) | 2 | 11
  Gefitinib: Day 1 of Cycle 1 | NA (NA) — Only 2 participants had evaluable Cmax at time point. For statistical reasons, calculation of summary statistics does not make sense for this low sample size. Individual values were 302 and 305 ng/mL. | 215 (48.7)
  Gefitinib: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 10
  Gefitinib: Day 15 of Cycle 1 | 432 (38.3) | 366 (32.6)

7. Secondary Outcome: Phase 1b: Average Observed Plasma Concentration (Cavg) of Tepotinib, Its Metabolites and Gefitinib
Description: Cavg is the average plasma concentration within 1 dosing interval obtained directly from the concentration versus time curve.
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 15 of Cycle 1 (each Cycle is 21 days)
Population: The PK analysis set employed here. "Number of participants analyzed" signifies participants who were evaluable for this outcome measure and "Number Analyzed" signifies those participants who were evaluable for specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 9
ng/mL
  Tepotinib | 654 (19.4) | 924 (43.3)
  MSC2571109A: number analyzed (Participants) | 6 | 8
  MSC2571109A | 185 (25.4) | 314 (52.6)
  MSC2571107A: number analyzed (Participants) | 6 | 8
  MSC2571107A | 36.4 (38.2) | 78.3 (76.0)
  Gefitinib | 321 (43.9) | 295 (29.0)

8. Secondary Outcome: Phase 1b: Minimum Observed Plasma Concentration (Cmin) of Tepotinib, Its Metabolites and Gefitinib
Description: Cmin is minimum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 9
ng/mL
  Tepotinib | 534 (18.8) | 735 (47.6)
  MSC2571109A: number analyzed (Participants) | 6 | 8
  MSC2571109A | 156 (28.8) | 270 (58.5)
  MSC2571107A: number analyzed (Participants) | 6 | 8
  MSC2571107A | 32.8 (40.1) | 68.7 (80.1)
  Geftinib | 231 (57.3) | 190 (43.5)

9. Secondary Outcome: Phase 1b: Time to Reach Maximum Plasma Concentration (Tmax) of Tepotinib, Its Metabolites and Gefitinib
Description: Tmax is time to reach maximum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 1 and 15 of Cycle 1 (each Cycle is 21 days)
Population: The Pharmacokinetic set included all participants who had received at least 1 dose of the tepotinib or gefitinib and who had provided at least 1 plasma concentration measurement of tepotinib or gefitinib after the first dose. Here "Number Analyzed" signifies those participants who were evaluable for specified category.
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Hours
  Tepotinib: Day 1 of Cycle 1: number analyzed (Participants) | 5 | 12
  Tepotinib: Day 1 of Cycle 1 | 8.00 [4.00 to 8.00] | 9.01 [4.00 to 10.00]
  Tepotinib: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 10
  Tepotinib: Day 15 of Cycle 1 | 6.00 [0.00 to 8.00] | 9.00 [4.00 to 24.00]
  MSC2571109A: Day 1 of Cycle 1: number analyzed (Participants) | 5 | 11
  MSC2571109A: Day 1 of Cycle 1 | 24.00 [23.75 to 24.00] | 24.00 [24.00 to 24.00]
  MSC2571109A: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 9
  MSC2571109A: Day 15 of Cycle 1 | 0.00 [0.00 to 24.00] | 0.00 [0.00 to 24.00]
  MSC2571107A: Day 1 of Cycle 1: number analyzed (Participants) | 5 | 11
  MSC2571107A: Day 1 of Cycle 1 | 24.00 [23.75 to 24.00] | 24.00 [24.00 to 24.00]
  MSC2571107A: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 9
  MSC2571107A: Day 15 of Cycle 1 | 0.13 [0.00 to 8.00] | 0.25 [0.00 to 24.00]
  Gefitinib: Day 1 of Cycle 1: number analyzed (Participants) | 2 | 11
  Gefitinib: Day 1 of Cycle 1 | NA [NA to NA] — Only 2 participants had evaluable tmax at time point. For statistical reasons, calculation of summary statistics does not make sense for this low sample size. Individual values were 4.00 and 4.00 hour. | 8.00 [4.00 to 8.02]
  Gefitinib: Day 15 of Cycle 1: number analyzed (Participants) | 6 | 10
  Gefitinib: Day 15 of Cycle 1 | 4.00 [4.00 to 10.00] | 8.00 [4.00 to 10.12]

10. Secondary Outcome: Phase 1b: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC 0-infinity) of Tepotinib, Its Metabolites and Gefitinib
Description: The AUC(0-inf) was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity.
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 1 and 15 of Cycle 1 (each Cycle is 21 days)
Population: The Pharmacokinetic set included all participants who had received at least 1 dose of the tepotinib or gefitinib and who had provided at least 1 plasma concentration measurement of tepotinib or gefitinib after the first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
ng*h/mL
  Tepotinib: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined.
  Tepotinib: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined.
  MSC2571109A: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined.
  MSC2571109A: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined.
  MSC2571107A: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined.
  MSC2571107A: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined.
  Gefitinib: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined.
  Gefitinib: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, AUC(0-inf) which is dependent on Lambda(z) was not determined.

11. Secondary Outcome: Phase 1b: Apparent Total Body Clearance From Plasma (CL/F) of Tepotinib and Gefitinib
Description: The CL/f is a measure of the rate at which it was metabolized or eliminated by normal biological processes. Clearance obtained after oral dose was influenced by the fraction of the dose absorbed. The CL/F from plasma was calculated using the formula: Dose divided by area under the concentration time curve from time zero to infinity (AUC0-inf).
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 15 of Cycle 1 (each Cycle is 21 days)
Population: The Pharmacokinetic set included all participants who had received at least 1 dose of the tepotinib or gefitinib and who had provided at least 1 plasma concentration measurement of tepotinib or gefitinib after the first dose. Here, "Number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 9
liter per hour (L/h)
  Tepotinib | 17.3 (19.6) | 20.3 (43.3)
  Gefitinib | 32.5 (44.1) | 35.3 (29.0)

12. Secondary Outcome: Phase 1b: Apparent Volume of Distribution (Vz/F) During the Terminal Phase of Tepotinib, Its Metabolites and Gefitinib
Description: The Vz/f was defined as the theoretical volume in which the total amount of required to uniformly distribute to produce the desired plasma concentration. Apparent volume of distribution after oral dose (Vz/F) was influenced by the fraction absorbed. The Vz/f was calculated by dividing the dose with area under the concentration time curve from time zero to infinity multiplied with terminal elimination rate constant Lambda(z). Vz/f=Dose/AUC(0-inf) multiply Lambda(z).
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 1 and 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Liter
  Tepotinib: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined.
  Tepotinib: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined.
  MSC2571109A: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined.
  MSC2571109A: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined.
  MSC2571107A: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined.
  MSC2571107A: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined.
  Gefitinib: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined.
  Gefitinib: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vz/F which is dependent on Lambda(z) was not determined.

13. Secondary Outcome: Phase 1b: Apparent Volume of Distribution During the Steady State (Vss/F) of Tepotinib, Its Metabolites and Gefitinib
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss/f after oral dose was influenced by the fraction absorbed.
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 1 and 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Liter
  Tepotinib: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined.
  Tepotinib: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined.
  MSC2571109A: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined.
  MSC2571109A: Day 15 of cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined.
  MSC2571107A: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined.
  MSC2571107A: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined.
  Gefitinib: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined.
  Gefitinib: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Vss/F which is dependent on Lambda(z) was not determined.

14. Secondary Outcome: Phase 1b: Apparent Terminal Elimination Rate Constant Lambda(z) of Tepotinib, Its Metabolites and Gefitinib
Description: Lambda(z) was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression method.
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 1 and 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1 per hour
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
1 per hour
  Tepotinib: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined.
  Tepotinib: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined.
  MSC2571109A: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined.
  MSC2571109A: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined.
  MSC2571107A: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined.
  MSC2571107A: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined.
  Gefitinib: Day 1 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined.
  Gefitinib: Day 15 of Cycle 1 | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined. | NA (NA) — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, Lambda (z) was not determined.

15. Secondary Outcome: Phase 1b: Apparent Terminal Half-Life (t1/2) of Tepotinib, Its Metabolites and Gefitinib
Description: Apparent terminal half-life was defined as the time required for the plasma concentration of drug to decrease 50 percent in the final stage of its elimination.
Time Frame: Pre dose, 0.25, 0.5, 1, 2, 4, 8, 10 and 24 hours post dose on Day 1 and 15 of Cycle 1 (each Cycle is 21 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Hours
  Tepotinib: Day 1 of Cycle 1 | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined. | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined.
  Tepotinib: Day 15 of Cycle 1 | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined. | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined.
  MSC2571109A: Day 1 of Cycle 1 | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined. | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined.
  MSC2571109A: Day 15 of Cycle 1 | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined. | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined.
  MSC2571107A: Day 1 of Cycle 1 | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined. | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined.
  MSC2571107A: Day 15 of Cycle 1 | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined. | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined.
  Gefitinib: Day 1 of Cycle 1 | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined. | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined.
  Gefitinib: Day 15 of Cycle 1 | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined. | NA [NA to NA] — Study drug administered once daily with rich PK sampling up to 24 hours. As half-life of study drug exceeding the PK sampling time, Lambda(z) could not be reliably estimated. Therefore, t1/2 which is dependent on Lambda(z) was not determined.

16. Secondary Outcome: Phase 1b: Percentage of Participants With Objective Response Based on Tumor Response Assessment According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) Criteria
Description: Objective response (OR) was defined as the percentage of participants who had achieved complete response (CR) or partial response (PR) as the best overall response according to local radiological assessments from randomization/the first administration of the study treatment to the first observation of disease progression (PD). CR: defined as disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR: defined as at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. PD defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Percentage of Participants | 33.3 [6.3 to 72.9] | 33.3 [12.3 to 60.9]

17. Secondary Outcome: Phase 1b: Percentage of Participants With Disease Control Based on Tumor Response Assessment According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) Criteria
Description: Disease control defined as CR, PR, or stable disease(SD) as the best overall response according to local radiological assessments from the date of randomization/the first administration of the study treatment to the first observation of PD. CR:disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR:at least 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. PD:an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5mm. SD:as any cases that do not qualify for either PR or PD at minimum interval of 42 days after randomization/start of study treatment
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Percentage of Participants | 50.0 [15.3 to 84.7] | 58.3 [31.5 to 81.9]

18. Secondary Outcome: Phase 1b: Number of Participants With Treatment-Related Treatment-Emergent Adverse Events (TEAEs) and Treatment-Related Serious TEAEs According to National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.03
Description: An adverse event (AE) was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Term TEAE was defined as AEs starting/worsening after first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs. Treatment-related AE was defined as having a "Possible" or "Related" relationship to study treatment, as assessed by the Investigator.
Time Frame: Up to 175 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Participants
  Any TEAE Related to Tepotinib | 6 | 9
  Any TEAE Related to Gefitinib | 5 | 11
  Any Serious TEAE Related to Tepotinib | 0 | 0
  Any Serious TEAE Related to Gefitinib | 0 | 0

19. Secondary Outcome: Phase 1b: Number of Participants With Grade 3/4 Treatment-Emergent Adverse Events (TEAEs) and Grade 3/4 Treatment-Related TEAEs According to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI-CTCAE) Version 4.03
Description: An adverse event (AE) was defined as any untoward medical occurrence in participant which does not necessarily have casual relationship with treatment was any unfavorable and unintended sign(including abnormal laboratory finding), symptom/disease temporally associated with use of medicinal product, whether/not considered related to medicinal product. Term TEAE was defined as AEs starting/worsening after first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs. Treatment-related TEAE was defined as having a "Possible" or "Related" relationship to study treatment, as assessed by the Investigator. As per NCI-CTCAE, Grade 3 is Severe, Grade 4 is Life-threatening and Grade 5 or Death. Number of participants with Grade 3/4 TEAEs and Grade 3/4 treatment-related TEAEs were reported.
Time Frame: Up to 175 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Participants
  Any Grade 3/4 TEAE | 5 | 9
  Any Grade 3/4 TEAE Related to Tepotinib | 2 | 4
  Any Grade 3/4 TEAE Related to Gefitinib | 0 | 0

20. Secondary Outcome: Phase 1b: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Leading to Permanent Treatment Discontinuation
Description: An adverse event (AE) was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Term TEAE is defined as AEs starting/worsening after first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs. Number of participants with TEAEs leading to permanent treatment discontinuation were reported.
Time Frame: Up to 175 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Participants
  TEAE Leading Permanent Tepotinib Discontinuation | 0 | 2
  TEAE Leading Permanent Gefitinib Discontinuation | 0 | 1

21. Secondary Outcome: Phase 1b: Number of Participants With Death and Reasons
Description: Number of participants with death due to progressive disease (PD), adverse event (AE) related to study treatment, AE not related to study treatment were reported. An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. PD defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 mm. Number of participants with deaths due to PD, AE related to study treatment, AE not related to study treatment were reported.
Time Frame: Up to 175 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Participants
  Death due to PD | 0 | 3
  Death due to AE related to study treatment | 0 | 0
  Death due to AE not related to study treatment | 1 | 0

22. Secondary Outcome: Phase 1b: Number of Participants With Laboratory Test Abnormalities of Grade 3 or Higher Severity Based on NCI-CTCAE Version 4.03 Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: The laboratory measurements included hematology and coagulation, biochemistry and urinalysis.
Time Frame: Up to 175 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Participants
  Amylase increased | 2 | 2
  Lipase increased | 1 | 2
  Neutrophil count decreased | 0 | 1
  Hyperglycemia | 0 | 2
  Hypocalcemia | 1 | 0
  Hyponatremia | 0 | 2
  Hypoproteinemia | 1 | 0

23. Secondary Outcome: Phase 1b: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs assessment included blood pressure, heart rate, respiratory rate and body temperature. Number of Participants with any clinically significant abnormalities in vital signs were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 175 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Participants | 0 | 0

24. Secondary Outcome: Phase 1b: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiograms (ECG) Findings
Description: ECG parameters included heart rhythm, pulse rate intervals, QRS, QT intervals, RR intervals and corrected QT(QTc) intervals. Clinical significance was determined by the investigator. Number of participants with clinically significant abnormalities in 12-lead ECG were reported.
Time Frame: Up to 175 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Participants | 0 | 0

25. Secondary Outcome: Phase 1b: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 2 or Higher Than 2
Description: ECOG PS score is widely used by doctors and researchers to assess how a participants' disease is progressing, and is used to assess how the disease affects the daily living abilities of the participant, and determine appropriate treatment and prognosis. The score ranges from Grade 0 to Grade 5, where Grade 0 = Fully active, able to carry on all pre-disease performance without restriction, Grade 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (like light house work, office work), Grade 2 = Ambulatory and capable of all self-care but unable to carry out any work activities, Grade 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours and Grade 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair, Grade 5 = Death. Number of participants with ECOG performance status score of 2 or higher than 2 were reported.
Time Frame: Up to 175 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg
Number analyzed (Participants) | 6 | 12
Participants | 1 | 9

26. Secondary Outcome: Phase 2: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Treatment-Related TEAEs and Treatment-Related Serious TEAEs According to National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.03
Description: An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs was defined as AEs that started or worsened in severity within the first dosing day of study treatment after the last dose of study treatment. TEAEs include both Serious TEAEs and non-serious TEAEs Treatment related AE was defined as having a "Possible" or "Related" relationship to study treatment, as assessed by the Investigator.
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 31 | 23 | 15
Participants
  Any TEAE | 31 | 23 | 13
  Any Treatment-Related TEAE | 30 | 23 | 11
  Any Serious TEAE | 13 | 8 | 5
  Any Treatment-Related Serious TEAE | 6 | 7 | 1

27. Secondary Outcome: Phase 2: Number of Participants With Greater Than or Equal to (>=) Grade 3 Treatment-Emergent Adverse Events (TEAEs) and >= Grade 3 Treatment-Related TEAEs According to National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.03
Description: An adverse event (AE) was defined as any untoward medical occurrence in participant which does not necessarily have casual relationship with treatment was any unfavorable and unintended sign(including abnormal laboratory finding), symptom/disease temporally associated with use of medicinal product, whether/not considered related to medicinal product. Term TEAE is defined as AEs starting/worsening after first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs. Treatment-related AE was defined as having a "Possible" or "Related" relationship to study treatment, as assessed by the Investigator. As per NCI-CTCAE, Grade 3 is Severe, Grade 4 is Life-threatening and Grade 5 or Death. Number of Participants With >= Grade 3 TEAEs and >= Grade 3 treatment-related TEAEs were reported.
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 31 | 23 | 15
Participants
  Any TEAE of >= Grade 3 | 20 | 14 | 7
  Any Treatment-related TEAE of >= Grade 3 | 16 | 12 | 1

28. Secondary Outcome: Phase 2: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Leading to Permanent Treatment Discontinuation
Description: as for outcome 20
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 31 | 23 | 15
Participants | 3 | 1 | 2

29. Secondary Outcome: Phase 2: Number of Participants With Death and Reasons
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. PD defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 mm. Number of participants with deaths due to progression disease (PD), AE related to study treatment, unknown reason was reported.
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 31 | 23 | 15
Participants
  Death due to disease progression | 21 | 15 | 8
  Death due to AE related to study treatment | 0 | 0 | 0
  Death due to unknown reason | 2 | 5 | 2

30. Secondary Outcome: Phase 2: Number of Participants With Laboratory Test Abnormalities of Grade 3 or Higher Severity Based on NCI-CTCAE Version 4.03 Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: The laboratory measurements included hematology and coagulation, biochemistry and urinalysis.
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 31 | 23 | 15
Participants
  Anaemia | 0 | 7 | 0
  Neutropenia | 0 | 1 | 0
  Alanine aminotransferase increased | 1 | 0 | 0
  Amylase increased | 7 | 2 | 2
  Gamma-glutamyltransferase increased | 0 | 1 | 0
  Lipase increased | 5 | 2 | 1
  Neutrophil count decreased | 2 | 3 | 0
  White blood cell count decreased | 1 | 2 | 0
  Hyponatremia | 1 | 3 | 0
  Hypokalemia | 0 | 2 | 0
  hypophosphatemia | 0 | 1 | 0
  Hypoalbuminemia | 1 | 0 | 0

31. Secondary Outcome: Phase 2: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: as for outcome 23
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 31 | 23 | 15
Participants | 0 | 0 | 0

32. Secondary Outcome: Phase 2: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiograms (ECG) Findings
Description: as for outcome 24
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 31 | 23 | 15
Participants | 2 | 1 | 0

33. Secondary Outcome: Phase 2: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 2 or Higher Than 2
Description: as for outcome 25
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 31 | 23 | 15
Participants | 6 | 1 | 1

34. Secondary Outcome: Phase 2 (Randomized Part Only): Progression-free Survival (PFS) Based on Tumor Assessment by Independent Review Committee (IRC)
Description: Progression-free survival (assessed by Independent Review Committee) time was defined as the time in months from randomization to either first observation of radiologically confirmed progression disease (PD) by the IRC or occurrence of death due to any cause within 84 days of either randomization or the last tumor assessment. PD is defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 mm. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Up to 328 weeks
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative)
Number analyzed (Participants) | 31 | 24
Months | 10.15 [4.24 to 19.32] | 4.34 [4.11 to 6.97]

35. Secondary Outcome: Phase 2: (Randomized Part Only): Overall Survival (OS) Time
Description: Overall survival time was measured as time in months between the date of randomization and the date of death.
Time Frame: Up to 328 weeks
Population: as for outcome 3
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative)
Number analyzed (Participants) | 31 | 24
Months | 17.25 [12.12 to 29.14] | 19.48 [15.90 to 21.82]

36. Secondary Outcome: Phase 2 (Randomized Part Only): Percentage of Participants With Objective Response Based on Tumor Response Assessment According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) Criteria
Description: as for outcome 16
Time Frame: Up to 328 weeks
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative)
Number analyzed (Participants) | 31 | 24
Percentage of Participants | 45.2 [29.7 to 61.3] | 33.3 [17.8 to 52.1]

37. Secondary Outcome: Phase 2 (Randomized Part Only): Percentage of Participants With Disease Control Based on Tumor Response Assessment According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) Criteria
Description: Disease control defined as CR, PR, or stable disease(SD) as the best overall response according to local radiological assessments from the date of randomization/the first administration of the study treatment to the first observation of PD. CR:disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR:at least 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. PD:an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5mm. SD:as any cases that do not qualify for either PR/PD at minimum interval of 42 days after randomization/start of study treatment.
Time Frame: Up to 328 weeks
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative)
Number analyzed (Participants) | 31 | 24
Percentage of Participants | 83.9 [69.0 to 93.4] | 70.8 [52.1 to 85.4]

38. Secondary Outcome: Phase 2 (Non-Randomized Part Only): Progression-free Survival (PFS) Based on Tumor Assessment by Investigator
Description: Progression-free survival (assessed by Investigator) time was defined as the time in months from randomization to either first observation of radiologically confirmed progression disease by the Investigator or occurrence of death due to any cause within 84 days of either randomization or the last tumor assessment. PD is defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 mm. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 15
Months | 1.41 [1.35 to 4.90]

39. Secondary Outcome: Phase 2 (Non-Randomized Part Only): Progression-free Survival (PFS) Based on Tumor Assessment by Independent Review Committee (IRC)
Description: Progression-free survival (assessed by Independent Review Committee) time was defined as the time in months from randomization to either first observation of radiologically confirmed progression disease by the IRC or occurrence of death due to any cause within 84 days of either randomization or the last tumor assessment. PD is defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study; and/or unequivocal progression of existing non-target lesions and/or the presence of new lesions. The sum must also demonstrate an absolute increase of at least 5 mm. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 15
Months | 2.63 [1.38 to 2.73]

40. Secondary Outcome: Phase 2: (Non-Randomized Part Only): Overall Survival (OS) Time
Description: Overall survival time was measured as time in months between the date of randomization and the date of death.
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 15
Months | 25.86 [13.08 to 39.66]

41. Secondary Outcome: Phase 2 (Non-Randomized Part Only): Percentage of Participants With Objective Response Based on Tumor Response Assessment According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) Criteria
Description: as for outcome 16
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 15
Percentage of Participants | 0 [0.0 to 18.1]

42. Secondary Outcome: Phase 2 (Non-Randomized Part Only): Percentage of Participants With Disease Control Based on Tumor Response Assessment According to Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST v1.1) Criteria
Description: as for outcome 37
Time Frame: Up to 328 weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 15
Percentage of Participants | 40 [19.1 to 64.0]

43. Secondary Outcome: Phase 2: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) Global Health Status Scale Score at End of Treatment (EOT)
Description: EORTC QLQ-C30 is a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. It consisted of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnoea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact. The EORTC QLQ-C30 GHS/QoL score ranges from 0 to 100; High score indicates better GHS/QoL. Score 0 represents: very poor physical condition and QoL. Score 100 represents: excellent overall physical condition and QoL.
Time Frame: Baseline and EOT (up to 110 weeks)
Population: Quality of life (Qol) evaluable population set included ITT participants in the treatment group in which they actually received the treatment with a baseline and at least 1 evaluable on-treatment QoL questionnaire. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 22 | 21 | 10
Units on a Scale | -16.29 (30.691) | -2.78 (22.869) | -24.19 (24.673)

44. Secondary Outcome: Phase 2: Time-to-Symptom Progression (TTSP)
Description: TTSP was measured from randomization to symptomatic progression by lung cancer symptom scale (LCSS) used to measure symptom changes relevant to quality of life (QoL).It consisted of 9 items focused on cancer symptoms (loss of appetite, fatigue, cough, shortness of breath, blood in sputum, pain, symptoms of cancer, illness affecting normal activity, QoL).For each symptom score distance from left boundary to point where participant has marked line was measured in millimeters (mm).Total scale length was 100 mm. Symptomatic progression was defined as increase/worsening of average symptomatic burden index (ASBI) (mean of 6 major lung cancer specific symptom scores);Worsening defined as 10% increase of scale breadth from baseline. Score 0 indicate no/minimum symptoms;100 indicates maximum level of symptoms.
Time Frame: Up to 328 weeks
Population: Quality of life (Qol) evaluable population set included ITT participants in the treatment group in which they actually received the treatment with a baseline and at least 1 evaluable on-treatment QoL questionnaire.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
Number analyzed (Participants) | 29 | 22 | 15
Months | 5.75 [1.41 to 11.86] | 7.95 [2.07 to 17.05] | 2.63 [1.41 to 8.31]

ADVERSE EVENTS:
Time Frame: Baseline up to 328 weeks
Description: The safety analysis set included all participants who had received any dose of the study medication.
Arm/Group | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) | Phase 2: Single-arm Cohort (MET+ T790M Positive)
All-Cause Mortality (participants affected / at risk) | 1/6 | 3/12 | 23/31 | 20/23 | 10/15
Serious Adverse Events (participants affected / at risk) | 4/6 | 7/12 | 13/31 | 8/23 | 5/15
Other Adverse Events (participants affected / at risk) | 6/6 | 12/12 | 31/31 | 23/23 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg (N=6) | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg (N=12) | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) (N=31) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) (N=23) | Phase 2: Single-arm Cohort (MET+ T790M Positive) (N=15)
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 2 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Face Oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 2 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Tepotinib 300 mg + Gefitinib 250 mg (N=6) | Phase 1b: Tepotinib 500 mg + Gefitinib 250 mg (N=12) | Phase 2: Tepotinib 500 mg + Gefitinib 250 mg (MET + T790 Negative) (N=31) | Phase 2: Pemetrexed and Cisplatin/Carboplatin (MET + T790 Negative) (N=23) | Phase 2: Single-arm Cohort (MET+ T790M Positive) (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 16 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 7 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0
Eyelids pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 4 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3 | 6 | 6 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 10 | 18 | 4 | 7
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 4 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 7 | 14 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 9 | 11 | 3
Asthenia (General disorders) | 1 | 0 | 5 | 5 | 2
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 2 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 6 | 1 | 1
Fatigue (General disorders) | 1 | 5 | 2 | 3 | 0
Malaise (General disorders) | 0 | 1 | 1 | 2 | 1
Oedema (General disorders) | 0 | 1 | 4 | 0 | 1
Oedema peripheral (General disorders) | 2 | 3 | 12 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 4 | 1 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 3 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 7 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 4 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 4 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 3 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 10 | 2 | 1
Amylase increased (Investigations) | 4 | 2 | 11 | 4 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 5 | 3 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 3 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 2 | 5 | 2
Blood creatinine increased (Investigations) | 2 | 0 | 4 | 6 | 2
Blood urea increased (Investigations) | 0 | 0 | 0 | 3 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 2 | 0 | 3 | 3 | 1
Electrocardiogram QT prolonged (Investigations) | 3 | 1 | 3 | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 4 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 2 | 1 | 1
International normalised ratio increased (Investigations) | 3 | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 2 | 2 | 8 | 3 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 2 | 9 | 1
Platelet count decreased (Investigations) | 1 | 0 | 2 | 6 | 0
Prothrombin time prolonged (Investigations) | 3 | 0 | 1 | 2 | 1
Weight decreased (Investigations) | 0 | 3 | 6 | 6 | 3
White blood cell count decreased (Investigations) | 1 | 0 | 2 | 12 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4 | 11 | 10 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 9 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 6 | 3 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 6 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 3 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 | 0 | 3 | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 3 | 4 | 0
Headache (Nervous system disorders) | 0 | 1 | 7 | 3 | 0
Innsomnia (Psychiatric disorders) | 1 | 1 | 5 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 8 | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 8 | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 3 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 4 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 8 | 0 | 4
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Inadequate diet (Social circumstances) | 0 | 0 | 1 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Bacterial test positive (Investigations) | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 0 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac discomfort (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT01982955/Prot_001.pdf
  • Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT01982955/SAP_000.pdf